CLINICAL TRIAL: NCT04355871
Title: Characteristics and Predictors of Death Among Hospitalized Patients With COVID-19 in Spain
Brief Title: Characteristics and Outcomes of Hospitalized Patients With COVID-19 in Spain
Acronym: COVID19@Spain
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19/SEIMC-FSG
Record Dates: First submitted 2020-04-19; First posted 2020-04-21 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2020-04

CONDITIONS: Covid19
Keywords: Covid19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19@Spain is a retrospective cohort study that aims to determine the clinical characteristics of hospitalized patients with COVID-19 in Spain and to identify prognostic factors of mortality and the need for mechanical ventilation

DETAILED DESCRIPTION:
COVID-19@Spain is a retrospective cohort study of patients admitted to Spanish hospitals with laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

The Ethics Committee for Research with Medicines of Hospital General Universitario Gregorio Marañón approved the study and waived informed consent for the collection of clinical data.

Investigators from participating centers were asked to include the first consecutive hospitalized patients (up to 100) meeting the study criteria from the start of the epidemic until March 17, 2020.

The data source was the electronic medical records. All data were entered directly by personnel at each institution using an online case report form (CRF), that satisfied local requirements of data confidentiality.

The variables registered included administrative data, epidemiological information, type of clinical specimen in which the diagnosis was confirmed, and the RT-PCR cycle threshold (Ct) of the confirmatory gene. We also registered demographics, comorbidities and current medications, signs and symptoms at admission, baseline laboratory tests results, chest X-ray findings at baseline and during follow-up, complications during hospitalization, medications with potential activity against COVID-19, and supportive treatments including oxygen therapy, admission to intensive care unit (ICU), mechanical ventilation (intubation), and use of adjuvant anti-inflammatory medications such as tocilizumab and systemic corticosteroids. Drug-related adverse events of medications for COVID-19 needing discontinuation were also recorded. The clinical status of the patients as of April 17, 2020, was categorized as discharged alive (with the date of discharge), alive and currently hospitalized, and death (with the date of death).

The primary endpoint is all-cause mortality at day 28, and the secondary endpoint is the need for mechanical ventilation. Baseline was the date of hospital admission. The follow-up censoring date is April 17, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay
* Hospital admission

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Spanish hospitals with laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Investigators from participating centers were asked to include the first consecutive hospitalized patients (up to 100) meeting the study criteria from the start of the epidemic until March 17, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4035 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 28 days

SECONDARY OUTCOMES:
Mechanical ventilation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ramón Arribas, MD, Principal Investigator — H. Univ. La Paz; Juan Berenguer, MD, Principal Investigator — H. Univ. Gregorio Marañón; Pablo Ryan, MD, Principal Investigator — H. Univ. Infanta Leonor; Jesús Rodriguez Baños, MD, Principal Investigator — H. Univ. Virgen Macarena; Jordi Carratala, MD, Principal Investigator — H. Univ. de Bellvitge; Jerónimo Pachón, MD, Principal Investigator — H. Univ. VIrgen del Rocio
Locations (128):
- Spain (128):
  - Comp. Hosp. Univ. A Coruña, A Coruña
  - H. Quiron A Coruña, A Coruña
  - H. de Alcaniz, Alcañiz
  - H. Gral Univ. de Alicante, Alicante
  - H. Univ. San Juan de Alicante, Alicante
  - H. Univ. de la Ribera, Alzira
  - H. Santos Reyes, Aranda de Duero
  - Hospital Alto Deba, Arrasate / Mondragón
  - H. Dr. Jose Molina Orosa, Arrecife
  - Complejo Asistencial de Avila, Ávila
  - Consorcio Sanitari Integral (CAIDM), Barcelona
  - H. Clinic, Barcelona
  - H. del Mar, Barcelona
  - H. Parc Sanitari Sant Joan de Deu, Barcelona
  - H. Santa Creu y Sant Pau, Barcelona
  - H. Univ. de Bellvitge, Barcelona
  - H. Vall d'Hebron, Barcelona
  - Hospital CIMA-Sanitas, Barcelona
  - SCIAS H. de Barcelona, Barcelona
  - H. Clinica de Benidorm, Benidorm
  - H. de Cruces, Bilbao
  - H. San Eloy_Barakaldo, Bilbao
  - H. Univ. de Basurto, Bilbao
  - H. Urduliz-Alfredo Espinosa, Bilbao
  - H. Gral de La Palma, Breña Alta
  - H. de Puerto Real, Cadiz
  - H. de Calahorra, Calahorra
  - H. Sant Jaume de Calella, Calella
  - H. Univ Santa Lucia, Cartagena
  - H. Univ de Henares, Coslada
  - Hospital Marina Salud de Dénia, Denia
  - Hospital Don Benito-Villanueva de la Serena, Don Benito
  - H. Gral Univ. de Elche, Elche
  - H. Univ. del Vinalopo, Elche
  - Comp. Hospt. Univ. de Ferrol, Ferrol
  - H. Francesc de Borja, Gandia
  - H. Comarcal de Blanes, Girona
  - H. de Figueres, Girona
  - H. Josep Trueta, Girona
  - H. Clinico San Cecilio, Granada
  - Hospital HLA Inmaculada, Granada
  - H. de Guadalajara, Guadalajara
  - H. de Guadarrama, Guadarrama
  - H. Juan Ramón Jiménez, Huelva
  - H. Riotinto, Huelva
  - H. Can Misses, Ibiza Town
  - H. Universitario de Jaén, Jaén
  - H. Univ. de Jerez de la Frontera, Jerez de la Frontera
  - H. Univ Insular de Gran Canaria, Las Palmas de Gran Canaria
  - H. Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - H. Univ. Severo Ochoa, Leganés
  - H. San Pedro, Logroño
  - H. Univ. Menez Rafael Mendez, Lorca
  - H. Lucus Augusti, Lugo
  - H. 12 de Octubre, Madrid
  - H. Clinica Univ. de Navarra_ Campus Madrid, Madrid
  - H. Clinico San Carlos, Madrid
  - H. Fundacion Jiménez Díaz, Madrid
  - H. Gral de la Defensa Gomez Ulla, Madrid
  - H. HLA Univ. Moncloa, Madrid
  - H. HM Sanchinarro, Madrid
  - H. Puerta de Hierro, Madrid
  - H. Univ HM Madrid, Madrid
  - H. Univ Principe de Asturias, Madrid
  - H. Univ. de Alcorcón, Madrid
  - H. Univ. de Getafe, Madrid
  - H. Univ. de Móstoles, Madrid
  - H. Univ. Gregorio Marañon, Madrid
  - H. Univ. HM Monteprincipe, Madrid
  - H. UNiv. HM Puerta del Sur, Madrid
  - H. Univ. Infanta Leonor, Madrid
  - H. Univ. La Paz, Madrid
  - H. Univ. La Princesa, Madrid
  - H. Univ. Ramón y Cajal, Madrid
  - H. Univ. Rey Juan Carlos, Madrid
  - H. Costa del Sol, Marbella
  - H. de Mataro, Mataró
  - H. Marbella Internacional, Málaga
  - H. Virgen de la Victoria, Málaga
  - H. de Melilla, Melilla
  - H. de Mendaro, Mendaro
  - H. Virgen de la Arrixaca, Murcia
  - H. Vega Baja, Orihuela
  - H. Univ. Central de Asturias, Oviedo
  - H. de Palamos, Palamós
  - H. Son Espases, Palma de Mallorca
  - H. Son Llatzer, Palma de Mallorca
  - H. Clinica Univ. Navarra, Pamplona
  - H. Virgen del Puerto, Plasencia
  - H. El Bierzo, Ponferrada
  - H. Do Salnes, Pontevedra
  - H. UNiv. Los Arcos del Mar Menor, Pozo-Aledo
  - H. Santa Barbara, Puertollano
  - H. Parc Tauli, Sabadell
  - Complejo Asist. Univ. de Salamanca, Salamanca
  - H. de Donostia, San Sebastián
  - H. Infanta Sofia, San Sebastián de los Reyes
  - H. de l'Esperit Sant, Santa Coloma de Gramenet
  - H. U. de Canarias, Santa Cruz de Tenerife
  - H. Univ. Nuestra Sra. de la Candelaria, Santa Cruz de Tenerife
  - H. Univ. Marques de Valdecilla, Santander
  - H. Clinico Univ. Santiago de Compostela, Santiago de Compostela
  - H. Univ de Valme, Seville
  - H. Univ. Virgen del Rocio, Seville
  - H. Univ. Virgen Macarena, Seville
  - H. Virgen Macarena, Seville
  - H. Univ Joan XXIII, Tarragona
  - H. Mutua de Terrasa, Terrassa
  - Complejo Hospitalario Virgen de la Salud, Toledo
  - H. Univ. HM Torrelodones, Torrelodones
  - H. Quiron Salud Torrevieja, Torrevieja
  - H. Virgen de la Cinta, Tortosa
  - H. Reina Sofia de Tudela, Tudela
  - H. Arnau de Vilanova-Lliria, Valencia
  - H. Clinico Univ. de Valencia, Valencia
  - H. de Sagunto, Valencia
  - H. Univ. y Polit. La Fe, Valencia
  - H. Clin. Univ. de Valladolid, Valladolid
  - H. Rio Hortega, Valladolid
  - H. Alvaro Cunqueiro, Vigo
  - H. de Viladecans, Viladecans
  - H. de la Marina Baixa, Villajoyosa
  - Hospital de la Plana, Villarreal de Huerva
  - H. Univ de Alava, Vitoria-Gasteiz
  - H. Virgen de la Concha, Zamora
  - H. Lozano Blesa, Zaragoza
  - H. Miguel Servet, Zaragoza
  - H. Ntra. Sra. de Gracia, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided